CLINICAL TRIAL: NCT03146468
Title: Pilot Study of the Tolerability of Nivolumab for Relapsed or Residual Haematological Malignancies After Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Nivolumab for Relapsed or Residual Haematological Malignancies After Allogeneic Stem Cell Transplantation
Acronym: NIVALLO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMH 2016.281
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Haematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab treatment arm (Experimental): Nivolumab injection 3mg/kg intravenously every 2 weeks
  Interventions: Drug: Nivolumab Injection

INTERVENTIONS:
Drug: Nivolumab Injection — Human monoclonal antibody targeting programmed death-1 (PD-1) cell surface receptor
  Other Names: Opdivo

SUMMARY:
This is a prospective study of the safety and efficacy of nivolumab for the treatment of relapsed or residual haematological malignancies after allogeneic stem cell transplantation (alloSCT).

Eligible patients will receive nivolumab at a dose of 3mg/kg intravenously every 2 weeks. The primary objective is to evaluate the incidence, severity and treatment responsiveness of GVHD following nivolumab treatment post-alloSCT.

ELIGIBILITY:
Inclusion Criteria:

* Prior allogeneic stem cell transplant for a haematological malignancy
* Confirmed relapse of haematological malignancy or persistent disease post-alloSCT
* Immunosuppression cessation for minimum of 2 weeks
* Life expectancy > 2 months
* ECOG performance status 0-2
* Greater than or equal to 30% CD3+ donor chimerism
* Serum creatinine ≤ 1.5 times upper limit of normal OR creatinine clearance ≥ 40mL/min
* AST and ALT ≤ 3 times upper limit of normal
* Total bilirubin ≤ 1.5 times upper limit of normal (except patients with Gilbert Syndrome)
* Signed written informed consent

Exclusion Criteria:

* Current evidence of any grade of GVHD
* Prior history of grade 2 or higher acute GVHD
* Moderate chronic GVHD within the previous 6 months or any prior history of severe chronic GVHD
* Active, known or suspected autoimmune disease (excluding vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger)
* Positive hepatitis B virus surface antigen
* Positive hepatitis C virus antibody
* Known human immunodeficiency virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Graft versus host disease | 8 weeks
  Cumulative incidence of graft versus host disease
Graft versus host disease | 24 weeks
  Cumulative incidence of graft versus host disease
Graft versus host disease | 48 weeks
  Cumulative incidence of graft versus host disease

SECONDARY OUTCOMES:
Overall response rate | 8 weeks
  Complete remission and partial remission
Overall response rate | 16 weeks
  Complete remission and partial remission
Overall response rate | 24 weeks
  Complete remission and partial remission
Overall response rate | 48 weeks
  Complete remission and partial remission

CONTACTS AND LOCATIONS:
Overall Officials: David Ritchie, FRACP, PhD, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared by researchers outside of this clinical trial